CLINICAL TRIAL: NCT06046235
Title: Virtual Evaluations of Joint Health Using Wearable Sensors in Persons With Haemophilia (VESPA)
Acronym: VESPA
Status: Not yet recruiting | Type: Observational
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/HAEMO/01
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-02

CONDITIONS: Haemophilia
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent technological innovations have enabled the creation of portable and easy-to-wear sensors with incredible potential to alter the clinical practice of rehabilitation. Using wearable sensors we have gathered preliminary data in the clinical setting measuring walking ability and function. Preliminary data shows that these wearable sensors can detect improvements in walking ability and function after a 12-week physiotherapy exercise programme in boys with haemophilia. In this proposal, we want to test the use of these wearable sensors in the patient's home to remotely monitor joint health and the effects of rehabilitation for people with haemophilia. We expect that wearable sensor technology is an efficient and promising tool to evaluate and monitor joint health and pain in persons with haemophilia. If usable in the home setting, the wearable sensors have the potential to provide immediate real-time feedback on joint health and rehabilitation goals to the patient and their haemophilia care team without the patient having to leave their home. The project will also support educational activities with researchers and patients to ensure that the use of this new type of rehabilitation will be fully integrated with their future treatment and management.

DETAILED DESCRIPTION:
Haemophilia is a rare, inherited disease. Joint and muscle bleeding is the most common symptom, representing 80% of all bleeding episodes.6 Musculoskeletal bleeding triggers a degenerative process characterised by synovial hypertrophy, irreversible changes in the articular cartilage and bone and is the predominant clinical characteristic of the disorder.6 Disabling physical limitation and pain remain the main co-morbidities of haemophilia. One of the important issues for PWH is the availability of accurate information about their musculoskeletal health that enables them to make decisions about their treatment.

In the context of self-management and improvement of health, telemedicine and telerehabilitation is an attractive option in haemophilia to improve health status monitoring, treatment satisfaction and pain control management.1-2 In our recent systematic review7 we evaluated the measurement properties of performance-based methods used to evaluate physical function in cPWH. Multi-item clinical instruments scoring global musculoskeletal symptoms together with measurement of joint range of motion (ROM) were the most commonly used measures. Data on validity and test-retest repeatability were lacking together with studies of sufficient size. In 2018, Timmer et al.8 reviewed the measurement properties of tools developed to assess activities and participation in adults with haemophilia (aPWH). Of the five self-reported and four performance based measurement tools evaluated, methodological quality was limited owing to insufficient evaluation of measurement error, cross-cultural validity and responsiveness. At present, there is no consensus on a core outcome set for monitoring musculoskeletal and functional impact of haemophilia across the lifespan of the disease. The recently published guidelines on the management of haemophilia recommend assessment of body structure and function, as well as ability to participate in everyday tasks as important joint health outcomes.9 In our multi-centre study of 52 children aged 6-11 years we observed that despite normal clinical examinations and comparable levels of physical activity, young cPWH with a history of ankle joint haemorrhage had significantly reduced dynamic muscle strength together with atrophy of the knee extensors, ankle dorsi and plantarflexors when compared to age and size-matched typically developing peers.10-12 Utilising laboratory-based three-dimension motion capture wearable sensors, adaptations in walking were also found including greater knee flexion and ankle dorsiflexion motion, vertical ground reaction and knee flexion forces. When investigating relationships between muscle strength and motor performance we found that greater frequency of bleeds into the knee joint were associated with a reduced muscle strength of ankle plantarflexors, walking distance and ability to stand on one leg.13 Bleeding into the ankle joint was associated with reduced knee extensor strength. In addition, gait patterns were associated with negative performance of physical function and performance depended on muscle strength.7 Muscle weakness of the leg was strongly correlated to muscle atrophy, reduced walking distances, slower ascent/ descent of stairs, reduced ankle joint motion, greater knee flexion motion and forces at the knee and ankle joint during walking.

In aPWH, Lobet and colleagues found moderately strong relationships between ankle joint motion during walking and self-reported pain and stiffness.14 In aPWH, lower performance of timed up and go test, which involves standing from a chair, walking 3-metres, turning and returning to the chair and sitting down as a measure of lower limb strength and mobility, is linked with greater arthropathy.15 We recently completed a preliminary study of clinic-based wearable sensors in a randomised controlled trial to investigate the effects of a 12-week muscle strengthening intervention for boys with haemophilia. We found that the rehabilitation exercise programme improved walking ability, muscle strength and function in those randomised to the intervention when compared to the control group. Although underpowered due its focus on feasibility, the preliminary findings together with other studies suggest that the evaluation of physical and functional performance using wearable sensors might serve as a basis for clinical monitoring and predicting future bleeding and joint arthropathy in PWH.4-5 Questions remain regarding how to incorporate current clinical joint examinations, degree of arthropathy and physical capabilities into the optimal delivery of individualised prophylaxis to optimise outcomes for each patient, reduce the potential for continued joint damage, limit physical disability and improve quality of life.

Therapy involving rehabilitation programmes often require quantification of body movement to assess physical function and determine the effectiveness of an intervention. High quality collection of movement data requires gold-standard laboratory-based motion capture systems. However, these technical systems can only be used in controlled environments and require patients to visit clinics/laboratory for testing. With the current restrictions on clinical visits and the requirement for people to stay at home during the pandemic, an alternative approach to collecting movement data is required. Wearable sensors offer accurate measures of body movement (including physical function, gait analysis, and motor abilities) with portability to be used in patient's homes.16 At the Angelo Bianchi Bonomi Hemophilia and Thrombosis Centre, our colleagues in Milan who are co-applicants on this application recently trialled an exergame system using a WiiFit Barefoot and Xbox 360 camera to monitor rehabilitation efficacy and adherence in cPWH.17 Those boys using the exergames system reported high levels of satisfaction and engagement compared to those not using the exergames system. Additionally, physiotherapists reported greater ability to remotely supervise rehabilitation programmes.

Inertial measurement units (IMUs) are a type of wearable sensor that combine gyroscopic, magnetometer and accelerometer signals to define the orientation of limbs. When attached to limbs the orientation of two IMUs can be accurately tracked through intelligent data fusion algorithms to calculate joint motion angles during movement tasks. Using wearable IMU sensors we have gathered preliminary data in the clinical setting measuring walking ability and function. Preliminary data showed that these wearable sensors could detect improvements in walking ability and function after a 12-week physiotherapy exercise programme in boys with haemophilia.3-5 The psychometric properties, e.g. validity and reliability, of IMUs have been published demonstrating limb orientation and joint kinematics to be accurate and repeatable when compared to gold-standard lab-based technology. However, IMUs have not previously been applied in a home-care setting to monitor physical function in patients with haemophilia during a rehabilitation programme. If usable in the home setting the devices will enable immediate real-time feedback on joint health or rehabilitation goals to the patient and their haemophilia care team without the patient having to leave their home.

In comparison to motion capture, wearable sensors offer a viable alternative to track human movement. However, few studies have explored the ecological validity of using of IMUs in home-care environments. By comparing joint ROM and physical function measures from IMU devices in the clinic to the same measurement taken at home, this study will provide data on the feasibility of implementing wearable sensors to track health outcomes in haemophilia patients. Furthermore, the responsiveness of IMU measures will be assessed by tracking changes in ROM and physical functional during and following a physiotherapy exercise intervention. Such a system can assist the physiotherapist with monitoring a patient's progress remotely during rehabilitation as well as providing valuable feedback to the patient, thereby increasing the efficiency and effectiveness of the rehabilitation process and enable the optimal delivery of individualised treatment for persons with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe or moderate haemophilia (FVIII or FIX ≤ 5%)
* Aged > 12 years of age
* Inhibitor or non-inhibitor, previous or current

Exclusion Criteria:

* Diagnosis of mild haemophilia (FVIII or FIX > 5%)
* Diagnosis of von Willebrand Disease or other bleeding disorder
* Aged ≤ 12 years of age
* Participants requiring a sterile environment
* The use of an oxygen-rich environment at a participant's home
* Participants or another person at the participant's home, with sensitive medical equipment whose functions may be compromised by the introduction of the IMU units, such as a pacemaker or implantable defibrillator
* Bedridden patients
* Patients with severe cognitive or psychiatric disorders as confirmed by a medical diagnosis

Min Age: 13 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: adolescents (13-17 years of age) and adults with Diagnosis of severe or moderate haemophilia (FVIII or FIX ≤ 5%)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Knee and ankle joint range of motion using wearable Inertial Measurement Units (IMU) devices | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- EKHUFT, Canterbury, Kent, United Kingdom